CLINICAL TRIAL: NCT02446704
Title: Phase I/II Study of Olaparib and Temozolomide in Patients With Recurrent Small Cell Lung Cancer Following Failure of Prior Chemotherapy
Brief Title: Study of Olaparib and Temozolomide in Patients With Recurrent Small Cell Lung Cancer Following Failure of Prior Chemotherapy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zofia Piotrowska (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Zofia Piotrowska, Assistant Professor of Medicine, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-121
Record Dates: First submitted 2015-05-14; First posted 2015-05-18 (Estimated); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: Small Cell Lung Cancer
Keywords: Small Cell Lung Cancer; SCLC
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — olaparib; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Olaparib and Temozolomide (Experimental): - Dose escalation will occur using a standard 3+3 dose escalation approach, beginning in dose level I with dose cohorts and rules for escalation and de-escalation. Once the MTD is determined, the study will move to the phase II portion.
  * Olaparib- Oral, on determined days per cycle
  * Temozolomide- Oral, on determined days per cycle
  Interventions: Drug: Olaparib; Drug: Temozolomide

INTERVENTIONS:
Drug: Olaparib
  Other Names: Lynparza
Drug: Temozolomide
  Other Names: Temodar®

SUMMARY:
This research study is evaluating the combination of olaparib and temozolomide as a possible treatment for Small Cell Lung Cancer.

DETAILED DESCRIPTION:
This research study is a Phase I/II clinical trial, which has two parts. The participant will be asked to participate in one part of the study. The first part tests the safety of the combination of drugs and tries to define the appropriate dose to use for future studies. The second part tests whether the combination of drugs is effective in treating small cell lung cancer. "Investigational" means that the combination of drugs is being studied. It also means that the U.S. Food and Drug Administration (FDA) has not approved the combination of drugs for Small Cell Lung Cancer.

Olaparib (Lynparza) is FDA approved for the treatment of a type of ovarian cancer associated with a particular DNA change. Olaparib works by blocking the activity of a protein called poly (ADP-ribose) polymerase (PARP) which is involved in DNA repair. Cancer cells rely on PARP to repair their DNA and enable them to continue dividing. Olaparib has been used in research studies with other cancers. Information from those other research studies suggests that this drug may help to treat patients with small cell lung cancer. While it is not approved by the FDA for small cell lung cancer, it is considered part of standard treatment for other cancer.

Temozolomide (Temodar) is approved by the FDA for the treatment of a type of brain tumor, glioblastoma. It has been studied in small cell lung cancer in previous research studies. While it is not approved by the FDA for small cell lung cancer, it is considered part of standard treatment for relapsed disease.

In this research study, the investigators are looking for the maximum tolerated dose or MTD of the combination of olaparib and temozolomide that can be given safely. The investigators will also begin to collect information about the effects of the combination on small cell lung cancer

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet the following criteria on screening examination to be eligible to participate in the study. The eligibility criteria apply to both the phase I and phase II portions of the study.
* Participant must have histologically or cytologically confirmed small cell lung cancer and may not be a candidate for potentially curative therapy.
* Presence of measurable disease (RECIST 1.1): At least one lesion, not previously irradiated, that can be accurately measured at baseline as ≥ 10 mm in the longest diameter (except lymph nodes which must have short axis ≥ 15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI) and which is suitable for accurate repeated measurements.
* The small cell lung cancer must have progressed radiographically following a platinum-based (cisplatin and/or carboplatin) standard prior chemotherapy regimen. Any number of interval prior lines of therapy is allowed. Patients who have received prior platinum-based chemotherapy and radiation for limited stage SCLC and have subsequently developed relapsed disease are eligible, as long as the platinum-based therapy was given within 12 months prior to the time of relapse.
* Participant (male/female) must be ≥18 years of age.
* Participant must have normal organ and bone marrow function measured within 28 days prior to administration of study treatment as defined below:

  * Hemoglobin ≥ 10.0 g/dL
  * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
  * Platelet count ≥100 x 10^9/L
  * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN)
  * AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limit of normal (unless liver metastases are present in which case it must be ≤5 x ULN)
  * Serum creatinine ≤1.5 x institutional upper limit of normal (ULN)
* ECOG performance status 0-1
* Participant must have a life expectancy ≥ 16 weeks.
* Women of childbearing potential must have a negative urine or serum pregnancy test within 28 days of initial dose of olaparib and temozolomide AND must agree to the use of two highly effective forms of contraception (see Section 5.5) throughout their participation in the study and for at least 3 months after the last dose of olaparib and temozolomide, OR confirmed prior to treatment on day 1 to be postmenopausal or surgically sterile. Postmenopausal is defined as:

  * Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments,
  * LH and FSH levels in the post menopausal range for women under 50,
  * radiation-induced oophorectomy with last menses >1 year ago,
  * chemotherapy-induced menopause with >1 year interval since last menses, or surgical sterilisation (bilateral oophorectomy or hysterectomy).
* Participant is willing to comply with the protocol for the duration of the study, and undergo treatment and scheduled visits and examinations including follow up. Participant must obtain prior approval from insurance to reimburse for oral temozolomide for the duration of the study or agree to self-pay for oral temozolomide.

Exclusion Criteria:

* Participants who exhibit any of the following conditions at screening will not be eligible for admission into the study. The exclusion criteria apply to both the phase I and phase II portions of the study.
* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
* Previous enrollment in the present study.
* Participation in another clinical study with an investigational product during the 21 days prior to first dose of olaparib and temozolomide.
* Participants receiving any systemic chemotherapy, radiotherapy (except for palliative reasons), within 2 weeks from the last dose prior to study treatment (or a longer period depending on the defined characteristics of the agents used). The patient can receive a stable dose of bisphosphonates for bone metastases, before and during the study as long as these were started at least 4 weeks prior to treatment with olaparib and temozolomide.
* Participants are to discontinue the use of the following classes of inhibitors of CYP3A4. Patients who are on these drugs are eligible if a washout period of a minimum of 7 days occurs before start of olaparib and temozolomide.

  * Azole antifungals
  * Macrolide antibiotics
  * Protease inhibitors
* Persistent clinically significant toxicities (>=CTCAE v. 4.0 grade 2) caused by previous cancer therapy, with the exception of alopecia.
* Participants with a previously documented diagnosis of myelodysplastic syndrome (MDS) (or any dysplastic leukocyte morphology suggestive of MDS) or acute myeloid leukaemia.
* Participants with symptomatic uncontrolled brain metastases. Baseline brain imaging by CT or MRI is required for all patients. Participants with brain metastases that have been treated with prior radiation therapy and are stable on a subsequent scan are allowed. Participants with untreated possible brain metastases that are new at the time of screening and are < 1 cm and asymptomatic are allowed. The participant can receive corticosteroids as long as these were started and at a stable dose at least 28 days prior to treatment.
* Major surgery within 14 days of starting study treatment and patients must have recovered from any effects of any major surgery.
* Participants considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, QTc prolongation > 470 msec, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, unstable spinal cord compression (untreated and unstable for at least 28 days prior to study entry), extensive bilateral lung disease with less than 20% predicted lung function by DLCO (Lung Diffusion Capacity Testing), or any psychiatric disorder that prohibits obtaining informed consent.
* Participants unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
* Pregnant or Breast feeding women. All patients (male and female) must agree to practice a medically acceptable method of contraception as defined in section 5.5. Should a woman become pregnant or suspect that she is pregnant while participating in this study, she should inform her treating physician immediately.
* Patients who have a history of and are known to be serologically positive for human immunodeficiency virus (HIV) and are receiving antiviral therapy. Baseline testing is not required.
* Patients with known active Hepatitis B or C. Baseline testing is not required.
* Patients with a known hypersensitivity to olaparib or any of the excipients of the product.
* Patients with uncontrolled seizures.
* Patients with second primary cancer, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumors curatively treated with no evidence of disease for ≥ 5 years.
* Patients with current and symptomatic pneumonitis, or extensive bilateral lung disease on high resolution CT scan.
* Patients with whole blood transfusion in the last 120 days prior to entry to the study.
* Patients with previous allogeneic bone marrow transplant.
* Patients with active, uncontrolled infection.
* Patients who need to continue treatment with any prohibited medications listed in Section 5.6
* Patients who have not completed the appropriate washout period for the prohibited medications in Section 5.6

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-10-13 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
MTD of Olaparib and Temozolomide | 2 Years
  Primary outcome measure for Phase 1 portion
Overall Response Rate for Olaparib and Temozolomide | 2 Years
  Primary outcome measure for Phase 2 portion

SECONDARY OUTCOMES:
Safety, assessed using CTCAE version 4.0 criteria | 2 Years
Overall Survival | 2 Years
Progression Free Survival | 2 Years
Methylation promoter methylation status | 2 Years
PAR levels | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Anna Farago, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts